CLINICAL TRIAL: NCT04934930
Title: Adjustment of Chemotherapy Duration in Follicular Lymphoma Patients According to Peripheral Blood or Bone Marrow Minimal Residual Disease Status
Brief Title: Adjustment of Chemotherapy Duration in Follicular Lymphoma According to Minimal Residual Disease Status
Acronym: FLMRD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Rabin Medical Center (Other); Tel-Aviv Sourasky Medical Center (Other Government); Assuta Ashdod Hospital (Other); Ziv Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC-19-0209
Record Dates: First submitted 2021-04-08; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Prospective multicenter, single arm, phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reduced number of bendamustine cycles in patients with mid-induction MRD negativity (Experimental): Patients with follicular lymphoma treated with obinutuzumab bendamustine & achieving MRD negativity as well as complete metabolic response on PET-CT at mid-induction would continue obinutuzumab treatment while omitting bendamustin after 4 cycles.
  Interventions: Drug: Bendamustin; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Bendamustin — Chemotherapy
  Other Names: Ribomustin
Drug: Obinutuzumab — Immunotherapy
  Other Names: Gazyva

SUMMARY:
Follicular lymphoma (FL) is a chronic indolent malignancy, where treatment with 6 cycles of bendamustine obinutuzumab (BO) is highly effective but at a cost of increased adverse events.

Tumor specific DNA can be traced in blood and bone marrow of follicular lymphoma patients even after therapy, and when detected after lymphoma treatment it is referred to as minimal residual disease (MRD).

MRD elimination after effective lymphoma treatment is a marker for deep response and correlates with prolonged remission.

In this study we aim to omit chemotherapy after 4 cycles of treatment in patients achieving MRD elimination after 3 months of therapy, as well as complete metabolic response on positron emission computed tomography (PET-CT), hoping to preserve treatment effectiveness while reducing adverse events.

DETAILED DESCRIPTION:
Follicular lymphoma (FL) is the second most common type of non-Hodgkin's lymphoma, with an estimated incidence of 3.18 cases per 100000 people a year in the United States The disease is characterized by an indolent behavior, where often treatment is unnecessary at diagnosis, and a "watch & wait" approach is the standard of care for asymptomatic patients. FL is also a highly responsive disease for immuno-chemotherapeutic combinations, although most patients will eventually relapse. Since the disease is incurable & indolent in nature, the therapeutic strategy should aim for disease control, while using treatments with high safety profile in order to minimize the chance for life threatening adverse events.

Therapy with rituximab cyclophosphamide, doxorubicin, vincristine & prednisone (R-CHOP) combination & subsequent rituximab maintenance therapy for 24 months shows excellent results with a median progression free survival (PFS) of above a decade.

The more recent GALLIUM trial has shown that combining the monoclonal antibody obinutuzumab with chemotherapy is even more efficacious compared to rituximab combinations. When different combinations were examined in this trial the best results were achieved with the bendamustine-obinutuzumab (BO) combination with 3 year PFS of 84%. Unfortunately the trial also revealed a downside for this effective combination with higher rate of fatal adverse events among patients receiving 6 cycles of bendamustine combinations.

In patients with acute leukemia evaluation for minimal residual disease (MRD) is a routine procedure, and the nature & length of treatment are guided by MRD status at different time points during therapy.

Among FL patients treated with obinutuzumab-chemotherapy combinations, it has been shown that after 3 cycles of treatment about 90% of patients were MRD negative. In addition MRD negativity at the end of induction in either peripheral blood or bone marrow was found to be associated with improved outcomes in patients with 1st line treatment for FL as well as in the relapsed setting.

These findings raise the possibility for an MRD based treatment approach, where the duration of chemotherapy could be guided by MRD status at mid-induction. Eliminating chemotherapy while continuing immunotherapy after achievement of MRD negativity & complete metabolic remission on PET-CT at mid-induction could reduce treatment toxicity, while potentially preserving efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. FL grade I-IIIa, according to world health organization (WHO) classification, in patients who were not previously treated with chemotherapy, have a high tumor bulk & an indication for treatment, as defined by the Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria.
3. Eastern Cooperative Oncology Group (ECOG) performance status grade 0-2.
4. The presence of a molecular marker in bone marrow or peripheral blood for MRD assessment.

Exclusion Criteria:

1. FL grade IIIb.
2. HIV infection.
3. HBsAg positivity.
4. Active malignancy other than FL
5. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival among patients treated with 4 cycles of BO & 2 additional cycles of obinutuzumab. | Progression free survival will be assessed 24 months after the end of induction.
  Progression-free survival is defined as the time from randomization to the earliest event of progression, relapse, or death from any cause. progression-free survival, is assessed by the investigator.

SECONDARY OUTCOMES:
Progression of disease within 24 months (POD24) | POD24 will be assessed at 24 months after treatment initiation
  POD24 is defined as disease progression or death due to disease progression occurring within 24 months after treatment initiation, as assessed by the investigator.
Overall survival among patients treated with 4 cycles of BO & 2 additional cycles of obinutuzumab. | Overall survival will be assessed 24 months after the end of induction.
  Overall survival is defined as the time from study initiation to death from any cause.
The rate of MRD negativity persistence at 12 months among patients treated with 4 cycles of BO & 2 additional cycles of obinutuzumab. | Persistence of MRD negativity will be assessed 12 months after study initiation.
  MRD will be assessed at mid-induction, end of induction and subsequently every 6 months.
The proportion of adverse events among patients treated with 4 cycles of BO & 2 additional cycles of obinutuzumab. | The proportion of various adverse events will be assessed until 24 months from the end of induction.
  The proportion of various adverse events will be assessed as documented by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Uri Abadi, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medical center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No